CLINICAL TRIAL: NCT03402789
Title: Pilot Study to Evaluate Docosahexaenoic Acid as Treatment for Residual Amblyopia
Brief Title: Docosahexaenoic Acid (DHA) Supplementation in Amblyopia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Hopkins failed to review contract with company providing complimentary dha, support was withdrawn necessitating me to get more grant money to fund study which was unsucccessful.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00150865
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Amblyopia
Keywords: Docosahexaenoic acid; Long chain fatty acid
MeSH Terms: conditions — Amblyopia | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: single blinded randomized controlled pilot study with 2/3 of participants randomized into the treatment arm and 1/3 of participants randomized into the placebo arm.
Who Masked: Participant
Masking Description: The participants will not be informed of whether they are taking the treatment drug or the placebo. Technicians measuring participants' visual outcomes are also masked. The principal investigator and co-investigators will know how the patient's are randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Docosahexaenoic acid (DHA) arm (Experimental): Participants will receive a pill of docosahexaenoic acid 1,200mg daily in addition to 2 hours of daily eye patching of the affected eye.
  Interventions: Drug: Docosahexaenoic Acid
- Placebo arm (Placebo Comparator): Participants will receive a placebo pill daily in addition to 2 hours of daily eye patching of the affected eye.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Docosahexaenoic Acid — Docosahexaenoic acid 1,200mg daily plus 2 hours of eye patching daily
  Other Names: DHA
  Arms: Docosahexaenoic acid (DHA) arm
Drug: Placebo Oral Tablet — Placebo tablet daily plus 2 hours of eye patching daily
  Arms: Placebo arm

SUMMARY:
This study evaluates the addition of docosahexaenoic acid (DHA) to eye patching in the treatment of residual amblyopia in children ages 3 to 18 years old. Two thirds of participants will receive DHA along with eye patching, while one third of participants will receive a placebo along with eye patching.

DETAILED DESCRIPTION:
Amblyopia is the most common cause of monocular visual impairment in children and adults. There are well established therapies for this condition, which typically involve eye patching or atropine eye drops. Despite these therapies, a substantial proportion of treated patients have some degree of residual amblyopia, even when treatment takes place early during the critical period visual development.

Investigators have tried to augment standard amblyopia treatment with medications that appear to promote visual cortex plasticity, thus addressing the neuronal pathogenesis of amblyopia. For example, levodopa, was described as a possible drug to treat amblyopia due to its ability to enhance cortical plasticity. While the rationale behind such treatments is promising, results from well-powered clinical trials have not shown a statistically significant effect of these treatments.

Docosahexaenoic acid (DHA) is a long chain polyunsaturated fatty acid (LCPUFA) that is considered essential for the maturation of the developing brain and retina. DHA, which is commercially available a nutritional supplement, has been added to infant formula, with studies showing that it improves visual development in premature infants. Randomized studies have shown that DHA supplementation of infant formula results in higher visual acuity in infants. Our proposal is aimed at conducting a prospective randomized pilot study to provide a preliminary assessment of the efficacy and safety of DHA combined with daily ocular occlusion therapy in children and teenagers with residual amblyopia. To our knowledge, this would be the first study aiming to treat amblyopia with DHA. If found to be effective, DHA may be considered a safe and inexpensive adjunct to our conventional means of treating amblyopia.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 to < 18 years
* Amblyopia associated with strabismus, anisometropia, or both
* Visual acuity, measured in each eye (without cycloplegia) within 7 days prior to enrollment using letter matching or the ETDRS protocol as follows:

  * Visual acuity in the amblyopic eye of 20/50 to 20/400
  * Visual acuity in the sound eye of 20/25 or better
  * No improvement or decline in best-corrected amblyopic eye visual acuity between two consecutive visits at least 4 weeks apart using the same testing method and optimal spectacle correction (if needed), with no improvement of more than 4 letters or one logMAR line.
* Previous or current treatment of amblyopia with either patching or atropine drops
* Spectacle correction (if applicable) for measurement of enrollment visual acuity must meet the following criteria and be based on a cycloplegic refraction that is no more than 6 months old
* Ocular examination within 6 months prior to enrollment
* Parent available for at least 6 months of follow-up, has home phone (or access to phone), and willing to be contacted by clinical site staff
* In the investigator's judgment, the subject is likely to comply with prescribed treatment (e.g., no history of poor compliance with patching treatment).

Exclusion Criteria:

* Myopia more than -8.00 D (spherical equivalent) in either eye.
* Current vision therapy or orthoptics
* Ocular cause for reduced visual acuity
* Prior intraocular or refractive surgery
* Strabismus surgery planned within 6 months
* Known immunodeficiency or hypercoagulable state
* Known skin reactions to patch or bandage adhesives
* Current treatment with topical atropine
* Constant deviations larger than 35 prism diopters
* Patients whose guardians have significant language or hearing impairment that would inhibit them from understanding the consent form or the procedures of the study will be excluded

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual acuity response with DHA | 6 months
  Measurement of the visual acuity change in those in the DHA arm compared to the placebo arm

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Kraus, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Wilmer Eye Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pediatric Eye Disease Investigator Group; Repka MX, Kraker RT, Dean TW, Beck RW, Siatkowski RM, Holmes JM, Beauchamp CL, Golden RP, Miller AM, Verderber LC, Wallace DK. A randomized trial of levodopa as treatment for residual amblyopia in older children. Ophthalmology. 2015 May;122(5):874-81. doi: 10.1016/j.ophtha.2015.01.002. Epub 2015 Feb 9. PMID 25676904
- [Background] Moon K, Rao SC, Schulzke SM, Patole SK, Simmer K. Longchain polyunsaturated fatty acid supplementation in preterm infants. Cochrane Database Syst Rev. 2016 Dec 20;12(12):CD000375. doi: 10.1002/14651858.CD000375.pub5. PMID 27995607
- [Background] Simmer K. Long-chain polyunsaturated fatty acid supplementation in infants born at term. Cochrane Database Syst Rev. 2001;(4):CD000376. doi: 10.1002/14651858.CD000376. PMID 11687076
- [Background] Koletzko B, Cetin I, Brenna JT; Perinatal Lipid Intake Working Group; Child Health Foundation; Diabetic Pregnancy Study Group; European Association of Perinatal Medicine; European Association of Perinatal Medicine; European Society for Clinical Nutrition and Metabolism; European Society for Paediatric Gastroenterology, Hepatology and Nutrition, Committee on Nutrition; International Federation of Placenta Associations; International Society for the Study of Fatty Acids and Lipids. Dietary fat intakes for pregnant and lactating women. Br J Nutr. 2007 Nov;98(5):873-7. doi: 10.1017/S0007114507764747. Epub 2007 Aug 10. PMID 17688705
- [Background] Kuratko CN, Barrett EC, Nelson EB, Salem N Jr. The relationship of docosahexaenoic acid (DHA) with learning and behavior in healthy children: a review. Nutrients. 2013 Jul 19;5(7):2777-810. doi: 10.3390/nu5072777. PMID 23877090